CLINICAL TRIAL: NCT01251510
Title: Bile Acid-induced GLP-secretion. A Study in Cholecystectomized Subjects
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, David P. Sonne, MD, University Hospital, Gentofte, Copenhagen
Other Study IDs: GAL-INK I
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy adults
- Type 2 diabetes

SUMMARY:
PURPOSE

The goal of the present project is to unravel the importance of bile acid-induced GLP-1 secretion (via the G protein-coupled receptor TGR5) in human physiology.

In the present study the investigators examine the GLP-1 secretion in healthy subjects and cholecystectomised patients. Thereby the investigators aim to show, that cholecystectomised patients have reduced bileflow after a meal, and as a consequence exhibit a diminished GLP-1 response as compared to healthy subjects.

ELIGIBILITY:
Inclusion Criteria: (Healthy)

* Normal fasting plasma glucose
* Normal glucose tolerance
* Normal haemoglobin levels
* Informed content

Inclusion Criteria: (cholecystectomy group)

* Laparoscopic cholecystectomy <6 months. Indication: Gallstones.
* Normal fasting plasma glucose
* Normal glucose tolerance
* Normal haemoglobin levels
* Informed content

Exclusion Criteria: (both groups)

* Diabetes
* Pre diabetes (impaired glucose tolerance or impaired fasting glucose)
* 1st degree relatives with diabetes
* Obesity (BMI > 30)
* Inflammatory bowels disease
* Nephropathy
* Liver disease
* Medication which cannot be on hold for 24h

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects and cholcystectomised patients (chol)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
GLP-1 secretion | Postprandial

CONTACTS AND LOCATIONS:
Overall Officials: David P. Sonne, MD, Principal Investigator — Gentofte Hospital, University of Copenhagen
Locations (1):
- Gentofte University Hospital, Hellerup, Denmark

REFERENCES:
- [Derived] Sonne DP, Hare KJ, Martens P, Rehfeld JF, Holst JJ, Vilsboll T, Knop FK. Postprandial gut hormone responses and glucose metabolism in cholecystectomized patients. Am J Physiol Gastrointest Liver Physiol. 2013 Feb 15;304(4):G413-9. doi: 10.1152/ajpgi.00435.2012. Epub 2012 Dec 28. PMID 23275610